CLINICAL TRIAL: NCT04504630
Title: High-Definition Transcranial Direct Current Stimulation on Episodic Memory in Individuals With Amnestic Mild Cognitive Impairment and History of TBI
Brief Title: Noninvasive Brain Stimulation on Memory in Individuals With Mild Cognitive Impairment and History of Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Christian Lobue, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU-2019-1769; CDMRP-AZ190088 (Other Grant/Funding Number: CDMRP)
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Results first posted 2025-05-04 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Amnestic Mild Cognitive Impairment; Traumatic Brain Injury; Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active HD-tDCS (Active Comparator): Participants will receive 10 sessions of active stimulation (1 mA anodal HD-tDCS targeting dorsal anterior cingulate region for 20 minutes) across 2 weeks, with episodic memory tasks completed at baseline, immediate follow-up after session 10, and a 3-month follow-up.
  Interventions: Device: High Definition Transcranial Direct Current Stimulation
- Sham HD-tDCS (Sham Comparator): Participants will receive 10 sessions of sham stimulation across 2 weeks, with episodic memory tasks completed at baseline, immediate follow-up after session 10, and a 3-month follow-up.
  Interventions: Device: Sham HD-tDCS

INTERVENTIONS:
Device: High Definition Transcranial Direct Current Stimulation — This wireless device delivers a very low electrical current to focused regions on the scalp in order to modulate underlying brain circuits to promote neuroplasticity. The device will be fitted onto a neoprene EEG cap, with 1 anode electrode placed and surrounded by 4 cathode electrodes in a ring pattern. Electrical stimulation will be applied using a constant voltage cortical stimulator (Model D185, Digitimer Ltd, UK, maximal output 1000 V/1.5 A) with single square-wave 50-μs pulses (0.1 A/μs rise time).
  Arms: Active HD-tDCS
Device: Sham HD-tDCS — Sham HD-tDCS
  Arms: Sham HD-tDCS

SUMMARY:
The study will examine the efficacy of high definition transcranial direct current stimulation (HD-tDCS) and its influence on episodic memory in patients with amnestic mild cognitive impairment and a history of Traumatic brain injury. Ten sessions of HD-tDCS to the dorsal anterior cingulate region is expected to result in improvements in episodic memory measures immediately following the last session and at a 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 and older
* Native English speakers
* 12 years of education or higher
* Active diagnosis of aMCI
* History of TBI based on VA/DOD criteria

Exclusion Criteria:

* TBI within the past 2 years
* Lifetime history of stroke, transient ischemic attack, heart attack, or congestive heart failure
* Lifetime history of epilepsy
* Major psychiatric disorders (i.e., posttraumatic stress disorder, bipolar disorder, schizophrenia)
* Substance use disorder
* Has metal fragments in head
* Taking medications that may interact with the HD-tDCS effect (i.e., amphetamines, L-dopa, carbamazepine, sulpiride, pergolide, lorazepam, dextromethorphan, D-cycloserine, flunarizine, or ropinirole)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-12-05 (Actual); Primary Completion 2024-06-16 (Actual); Study Completion 2025-01-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to upload study data to the FITBIR repository system within one year of completion.

RESULTS

PARTICIPANT FLOW:
Groups:
- Active HD-tDCS: Participants will receive 10 sessions of active stimulation (1 mA anodal HD-tDCS targeting dorsal anterior cingulate region for 20 minutes) across 2 weeks.
- Sham HD-tDCS: Participants will receive 10 sessions of sham stimulation across 2 weeks.
Period: Assigned to Treatment
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Started | 18 | 8
Completed | 16 | 8
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: Started Treatment
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Started | 16 | 8
Completed | 16 | 8
Not Completed | 0 | 0
Period: Follow-Up at 3 Months
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Started | 16 | 8
Completed | 13 | 7
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active HD-tDCS | Sham HD-tDCS | Total
Number analyzed (Participants) | 16 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (5.6) | 72.5 (8.1) | 71.0 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 10 | 6 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 15 | 8 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 8 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 8 | 24
Time since diagnosis [Mean (Standard Deviation); unit: years] | 2.2 (1.8) | 1.5 (1.4) | 2.0 (1.7)
Education [Mean (Standard Deviation); unit: years] | 17.0 (2.2) | 17.4 (1.6) | 17.1 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Hopkins Verbal Learning Test-Revised Total Learning
Description: Episodic verbal memory will be assessed with the Hopkins Verbal Learning Test-Revised (HVLT-R). The HVLT-R is a verbal episodic memory task where a list of 12 words is read aloud for 3 consecutive trials followed by a 20 minute delayed recall trial. The number of items recalled immediately after each trial are summed to create a total learning score, ranging from 0-36. Also, the number of items recalled for the delayed trial are recorded as a delayed recall score, ranging from 0-12. Scores were converted to standardized scores (T-scores) using normative data, ranging from 2-86. Higher scores reflect better episodic memory performance.
Time Frame: Baseline, immediately following last HD-tDCS session, and again at 3-month follow-up
Population: 4 participants were lost to follow-up
Measure: Mean (Standard Deviation); unit: T-score on a scale
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 16 | 8
T-score on a scale
  Baseline | 35.8 (10.4) | 35.9 (8.0)
  Immediate Post-treatment | 34.2 (9.6) | 31.6 (4.4)
  3 Month Follow-up: number analyzed (Participants) | 13 | 7
  3 Month Follow-up | 32.7 (8.8) | 37.1 (17.2)

2. Primary Outcome: Hopkins Verbal Learning Test-Revised Delayed Recall
Description: as for outcome 1
Time Frame: Baseline, immediately following the last HD-tDCS session, and a 3-month follow-up
Population: 4 participants lost to follow-up
Measure: Mean (Standard Deviation); unit: T-score on a scale
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 16 | 8
T-score on a scale
  Baseline | 30.1 (12.8) | 31.0 (14.1)
  Immediate Post-treatment | 27.7 (11.4) | 26.9 (8.2)
  3-Month Follow-up: number analyzed (Participants) | 13 | 7
  3-Month Follow-up | 26.9 (10.5) | 32.4 (17.9)

3. Primary Outcome: Brief Visuospatial Memory Test-Revised (BVMT-R) Total Learning
Description: Episodic verbal memory will be assessed with the Brief Visuospatial Memory Test-Revised (BVMT-R). The BVMT-R is a visual episodic memory task where where an array of 6 simple geometric visual designs are presented in a 2 x 3 matrix for 10 seconds for 3 trials. The number of items recalled immediately after each trial are summed for accuracy and placement to create a total learning score, ranging from 0-36. Also, the number of items recalled for the delayed trial are recorded as a delayed recall score, ranging from 0-12. Scores were converted to standardized scores (T-scores) using normative data, ranging from 2-86. Higher scores reflect better episodic memory performance.
Time Frame: Baseline, immediately post-treatment, and a 3 -month follow-up
Population: 1 participant in active HD-tDCS group did not complete the BVMT-R immediately post-treatment. 4 participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: T-score on a scale
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 16 | 8
T-score on a scale
  Baseline | 33.0 (10.0) | 29.1 (8.9)
  Immediate Post-treatment: number analyzed (Participants) | 15 | 8
  Immediate Post-treatment | 32.3 (10.4) | 33.3 (7.0)
  3-Month Follow-up: number analyzed (Participants) | 13 | 7
  3-Month Follow-up | 33.8 (8.1) | 34.1 (12.0)

4. Primary Outcome: Brief Visuospatial Memory Test-Revised Delayed Recall
Description: as for outcome 3
Time Frame: Baseline, immediately post-treatment, and a 3-month follow-up
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: T-score on a scale
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 16 | 8
T-score on a scale
  Baseline | 32.6 (9.8) | 32.4 (9.4)
  Immediate Post-treatment: number analyzed (Participants) | 15 | 8
  Immediate Post-treatment | 32.4 (11.9) | 32.0 (8.6)
  3-Month Follow-up: number analyzed (Participants) | 13 | 7
  3-Month Follow-up | 31.6 (12.9) | 32.4 (11.1)

5. Secondary Outcome: Phonemic Fluency
Description: The phonemic verbal fluency task is a measure of language. The subject is required to name as many words as possible that begin with specified letters within 1 minute. Three different letter trials are completed. The outcome measure for this task is the total number of correct responses across the trials, ranging from 0-90. Scores were converted to standardized scores (T-scores) using normative data, ranging from 2-86. Higher scores reflect better performance.
Time Frame: Baseline, immediately post-treatment, and a 3-month follow-up
Population: 4 participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: T-score on a scale
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 16 | 8
T-score on a scale
  Baseline | 45.8 (9.1) | 49.1 (13.9)
  Immediately Post-treatment | 46.3 (5.8) | 53.0 (14.1)
  3-Month Follow-up: number analyzed (Participants) | 13 | 7
  3-Month Follow-up | 49.1 (8.1) | 54.6 (13.9)

6. Secondary Outcome: Semantic Fluency
Description: The semantic verbal fluency task is a measure of language and involves 3 conditions. The subject is required to name as many animals as possible within 1 minute. The outcome measure for this task is the total number of correct responses, ranging from 0-90. Scores were converted to standardized scores (T-scores) using normative data, ranging from 2-86. Higher scores reflect better performance.
Time Frame: Baseline, immediate post-treatment, and a 3-month follow-up
Population: 4 participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: T-score on a scale
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 16 | 8
T-score on a scale
  Baseline | 38.4 (14.7) | 37.4 (15.4)
  Immediate Post-treatment | 38.6 (16.3) | 42.2 (17.8)
  3-Month Follow-up: number analyzed (Participants) | 13 | 7
  3-Month Follow-up | 37.3 (13.8) | 38.4 (18.2)

7. Secondary Outcome: Trail Making Test
Description: The Trail Making Test is a measure of cognitive flexibility and executive functions. The task requires the subject to as quickly as possible complete two conditions, involving number sequencing and then number-letter switching. The outcome measure for this task is the time in seconds to complete the number-letter switching condition, ranging from 15-300. Scores were converted to standardized scores (T-scores) using normative data, ranging from 2-86. Higher scores reflect better performance
Time Frame: Baseline, immediate post-treatment, and a 3-month follow-up
Population: 4 participants were lost to follow-up
Measure: Mean (Standard Deviation); unit: T-score on a scale
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 16 | 8
T-score on a scale
  Baseline | 41.6 (15.9) | 41.9 (13.3)
  Immediate Post-treatment | 45.7 (10.2) | 44.1 (16.4)
  3-Month Follow-up: number analyzed (Participants) | 13 | 7
  3-Month Follow-up | 47.8 (17.6) | 39.1 (20.1)

8. Secondary Outcome: Stroop Color and Word Test
Description: The Stroop Color and Word Test is a measure of information processing speed and complex attention. The task requires the subject to as quickly as possible complete 3 conditions, involving word reading, color naming, and response inhibition. The outcome measure for this task was the response inhibition trial, which is scored as the total correct items completed in the administration time of 45 seconds, ranging from 0-100. Scores were converted to standardized scores (T-scores) using normative data, ranging from 2-86. Higher scores reflect better performance.
Time Frame: Baseline, immediate post-treatment, and a 3-month follow-up
Population: 4 participants were lost to follow-up
Measure: Mean (Standard Deviation); unit: T-score on a scale
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 16 | 8
T-score on a scale
  Baseline | 38.8 (6.9) | 39.1 (10.3)
  Immediate Post-treatment | 41.6 (9.8) | 40.0 (9.6)
  3-Month Follow-up: number analyzed (Participants) | 13 | 7
  3-Month Follow-up | 39.9 (12.4) | 37.9 (11.8)

9. Secondary Outcome: Digit Span Test
Description: The Wechsler Adult Intelligence Scale-4 Digit Span Test measures simple attention and working memory. The examiner reads aloud a series of numbers of increasing length, and individuals are required to repeat each series across 3 separate conditions, involving forwards, backwards, and in sequence. Each trial is scored as incorrect (0) or correct (1), and the total number of correct trials across the 3 conditions are summed, ranging from 0-48. Scores were converted to standardized scores (scaled-scores) using normative data, ranging from 1-19. Higher scores reflect better episodic memory performance
Time Frame: Baseline, immediate post-treatment, and a 3-month follow-up
Population: 1 participant did not complete the Digit Span Test in the active HD-tDCS group at the 3-month follow-up. 4 participants were lost to follow-up.
Measure: Mean (Standard Deviation); unit: Scaled score on a scale
Arm/Group | Active HD-tDCS | Sham HD-tDCS
Number analyzed (Participants) | 16 | 8
Scaled score on a scale
  Baseline | 10.8 (2.0) | 9.8 (1.8)
  Immediate Post-treatment | 10.6 (1.7) | 10.4 (1.8)
  3-Month Follow-up: number analyzed (Participants) | 12 | 7
  3-Month Follow-up | 10.8 (2.0) | 9.4 (2.1)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the start of assigned treatments (1 mA and sham) through study completion. This involved collection of information about adverse effects daily at the beginning and end of each treatment session and then again at the 3-month follow-up visit.
Arm/Group | Active HD-tDCS | Sham HD-tDCS
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/8
Other Adverse Events (participants affected / at risk) | 0/16 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active HD-tDCS (N=16) | Sham HD-tDCS (N=8)
Nausea and Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT04504630/Prot_SAP_001.pdf
  • Informed Consent Form (2023-09-11): https://cdn.clinicaltrials.gov/large-docs/30/NCT04504630/ICF_000.pdf